CLINICAL TRIAL: NCT01816022
Title: Myeloproliferative Neoplasms and Bone Structure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Sarah Farmer, MD, University of Southern Denmark
Other Study IDs: HFEX 11.15
Record Dates: First submitted 2012-09-18; First posted 2013-03-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis
Keywords: CMPN; Fracture; Osteoporosis; Biochemical Bone Markers
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Fractures, Bone; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples to compare groups and to look for endocrine abnormalities
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a clinical study to evaluate the effect of CMPN (Chronic myeloproliferative neoplasm) to the bone.

The hypothesis is that patients with CMPN have a higher fracture-rate compared to the background population. We expect to find a lower BMD using conventional DXA scan (dual energy x-ray absorptiometry), and a change in other parameters using HR-pQCT (high-resolution peripheral quantitative computerized tomography).Biochemical bone markers is measured to support the hypothesis.

DETAILED DESCRIPTION:
This is a clinical study to evaluate the effect of CMPN to the bone.

Three individual cohorts are defined; a cohort consisting of 50 patients with Polycythemia Vera (PV), a cohort consisting of 50 patients with Essential Thrombocythemia (ET), and a cohort consisting of 25 patients with Primary Myelofibrosis (PMF).

Patients are recruited from the Department of Hematology, Odense University Hospital.

Interventions consist of:

* Conventional DXA scan to measure Bone Mineral Density (BMD).
* Experimental HR-pQCT to assess geometry, strength and microstructure of the bone in 3 dimension.
* Blood-samples are collected and frozen for later analyses of Biochemical Bone Markers: 1-CTP, Ctx, ALP (alkaline phosphatase)and P1NP.

The outcome is compared to healthy control individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PV (according to WHO 2008 criteria), only JAK2-pos.(Janus kinase 2)
* Diagnosis of ET (according to WHO 2008 criteria), only JAK2-pos.
* Diagnosis of PMF (according to WHO 2008 criteria)independent of JAK2-status.

Exclusion Criteria:

* Pregnancy
* Bone Diseases (Mb. Pagets, Myelomatosis, MGUS (monoclonal gammopathy of undetermined significance), osteogenesis imperfecta, Prim. hyperparathyroidism, osteomalacia.
* Drugs (Prednisone>3 mth, anti-osteoporotic drugs, anti-estrogen drugs.
* Presence of any psychologic condition or language barrier, which may interfere which a complete understanding, and arise ethnical considerations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Danish patients with CMPN
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | 1 day
  Patients will undergo one DXA scan independent of time of CMPN diagnosis

SECONDARY OUTCOMES:
Evaluation of Geometry, Strength and Micro-Structure of the bone. | 1 day
  Patients will undergo one HR.pQCT indepedent of the time of the diagnosis of CMPN

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Farmer, MD, Principal Investigator — Department of Hematology, Clinical Institute, University of Southern Denmark
Locations (1):
- Faculty of Health Sciences, Institute of Clinical Research, Odense, Region Syddanmark, Denmark

REFERENCES:
- [Derived] Farmer S, Vestergaard H, Hansen S, Shanbhogue VV, Stahlberg CI, Hermann AP, Frederiksen H. Bone geometry, bone mineral density, and micro-architecture in patients with myelofibrosis: a cross-sectional study using DXA, HR-pQCT, and bone turnover markers. Int J Hematol. 2015 Jul;102(1):67-75. doi: 10.1007/s12185-015-1803-3. Epub 2015 May 5. PMID 25939704